CLINICAL TRIAL: NCT04663048
Title: Evaluation of a Reduced Photorefractive Intrastromal Corneal Crosslinking Illumination Protocol. A Randomized Controlled Trial.
Brief Title: PiXL as a Treatment for Low Grade Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PiXLMYOP-III
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Myopia; Refractive Errors
Keywords: Corneal Crosslinking
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants are not aware which eye will receive the reduced treatment and which eye will receive the ordinary treatment time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol A (Experimental): PiXL treatment with pulsed UV illumination (1.0 sec on /0.8 sec off) in high oxygen in a central ring-shaped 3.5-mm zone of the cornea and total illumination time of 10 min. The area consist of three rings with a central 1.5-mm zone that is left untreated. The illumination area consists of three rings, where the outer and inner ring are thinner than the middle ring. The maximum energy is distributed in the middle ring.
  Interventions: Procedure: PiXL
- Protocol B (Active Comparator): PiXL treatment with pulsed (0.5 sec on / 1 sec off) UV illumination in high oxygen in a central ring-shaped 3.5-mm zone of the cornea and total illumination time of 16:40 min. The area consist of three rings with a central 1.5-mm zone that is left untreated. The illumination area consists of three rings, where the outer and inner ring are thinner than the middle ring. The maximum energy is distributed in the middle ring.
  Interventions: Procedure: PiXL

INTERVENTIONS:
Procedure: PiXL — Phototherapeutic intrastromal corneal collagen cross-linking (PiXL) performed in a high-oxygen environment without corneal epithelial debridement, for treatment of low grade myopia.

SUMMARY:
To assess the improvement in myopia with phototherapeutic intrastromal corneal collagen cross-linking (PiXL) without epithelial debridement (epi-on) in high oxygen environment for low grade myopia. The study compares two 3.5-mm central ring-shaped zone protocols; 10 min illumination time vs 16:40 min illumination time.

DETAILED DESCRIPTION:
The study design is a prospective, single-masked intraindividually comparing randomized controlled trial, conducted at the Department of Clinical Sciences / Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study includes healthy men and women with low grade myopia, aged between 18-35 years and involves 25 participants with a myopia of -0.50 to -2.5 diopters (D) and astigmatism of ≤0.75D. All participants are treated with phototherapeutic intrastromal corneal collagen cross-linking (PiXL) without epithelial debridement (epi-on), after topical riboflavin. Both eyes are treated and randomized to receive ultraviolet (UV) light according to PiXL Protocol A in one eye and PiXL Protocol B in the other, which is masked to the participant. Throughout the treatment, humidified oxygen is continuously delivered around the eye using an oxygen mask to achieve an oxygen concentration of ≥95 percentage. Prior to inclusion all participants are informed about the procedures and provide oral and written informed consent.

At baseline, each eye is examined with slit-lamp microscopy, subjective refraction, determination of uncorrected (UCVA), low contrast visual acuity at 2.5 percentage and 10 percentage contrast and best corrected (BSCVA) visual acuities using the LogMAR fast protocol and intraocular pressure (IOP) using Goldmann applanation tonometry. Under standardized, mesopic light conditions each eye is evaluated by keratometry readings, central corneal thickness and after treatment also the depth of demarcation lines, extracted from Schemipflug camera measurements, Pentacam HR® (Oculus, Inc. Lynnwood, WA). Central corneal endothelial photographs are taken with the Topcon SP-2000P specular microscope (Topcon Europe B.V., Capelle a/d Ijssel, the Netherlands), from which the corneal endothelial cell count is manually calculated from a cluster of 25 cells from each photograph. Total ocular wavefront is measured with iTrace (Tracey Technologies, Inc.).

All the above mentioned examinations are reassessed at 1, 3, 6 and 12 months after treatment. At 1 day and 1 week after treatment, solely UCVA, Auto refractor measurements, slit-lamp examination and a subjective comparison of discomfort and visual performance in each eye are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent on distance subjective refraction between -0.50D and -2.50D.
* Astigmatism ≤ 0.75D
* Stable myopia. Maximum change in refraction of 0.50D in the last 2 years.
* Best corrected visual acuity of at least 0.00 logMAR (ETDRS chart).
* Thinnest pachymetry reading ≥ 440 μm.
* No previous ocular surgery.
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* History of or current condition, disease, surgery or medication with ocular effects that could affect the outcomes of the treatment.
* Allergy to any substance or device used in the study.
* Cognitive insufficiency interfering with the informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-06-17 (Estimated); Study Completion 2024-06-17 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity (UDVA) | 1, 3, 6 and 12 months after treatment.
  Change from baseline in UDVA (logMAR)
Manifest Refractive Spherical Equivalent | 1, 3, 6 and 12 months after treatment
  Change from baseline in MRSE (Diopters)

SECONDARY OUTCOMES:
Best spectacle corrected visual acuity (BSCVA) | 1, 3, 6 and 12 months after treatment
  Change from baseline in BSCVA (logMAR)
Endothelial cell density (ECC) | 1, 3, 6 and 12 months after treatment
  Change from baseline in ECC (cells/mm^2)
Low contrast visual acuity at 10% and 2.5% (LCVA) | 1, 3, 6 and 12 months after treatment
  Change from baseline in LCVA 10 % and 2.5% (logMAR)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, MD, PhD, Principal Investigator — Umeå University Hospital
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No